CLINICAL TRIAL: NCT02975466
Title: Randomized Controlled Trial Comparing the Efficiency of Three Third Generation Supraglottic Airways as an Intubation Route
Brief Title: Comparing the Efficiency of Three Third-generation Supraglottic Airways as an Intubation Route
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Marie-Josee Colas, Anesthesiologist, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-1484
Record Dates: First submitted 2016-11-16; First posted 2016-11-29 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Difficult Intubation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AirQ Blocker supra-glottic airway device (Experimental): Group of patients in which the Air-Q Blocker will be used and measured as an intubation conduit.
  Interventions: Device: Insertion of AirQ Blocker and intubation through the device
- AuraGain supra-glottic airway device (Experimental): Group of patients in which the AuraGain will be used and measured as an intubation conduit.
  Interventions: Device: Insertion of AuraGain and intubation through the device
- I-Gel supra-glottic airway device (Experimental): Group of patients in which the I-Gel will be used and measured as an intubation conduit.
  Interventions: Device: Insertion of I-Gel and intubation through the device

INTERVENTIONS:
Device: Insertion of AirQ Blocker and intubation through the device — Insertion of the SGA device and evaluation of easiness of endotracheal intubation
  Arms: AirQ Blocker supra-glottic airway device
Device: Insertion of AuraGain and intubation through the device — Insertion of the SGA device and evaluation of easiness of endotracheal intubation
  Arms: AuraGain supra-glottic airway device
Device: Insertion of I-Gel and intubation through the device — Insertion of the SGA device and evaluation of easiness of endotracheal intubation
  Arms: I-Gel supra-glottic airway device

SUMMARY:
A "can't intubate, can't oxygenate" situation is life-threatening and the physician must be prepared to react quickly. Similarly, a difficult intubation with adequate ventilation is associated with complications. In both of these situation and as recommend by different societies, a supra-glottic airway (SGA) device can be used to help ventilation, or as an intubation conduit to ease the airway access. The objective of this randomized controlled trial is to establish which SGA, between the AuraGain, AirQ Blocker and I-Gel, allows the fastest intubation time in an adult population, with the objective of minimizing complications related to these situations. The investigators will conduct a three-arm trial to compare different outcomes related to the installation of the SGA and its use as an intubation conduit. The results of this trial will inform the anesthesiologist on which device to use on to have close in case of airway emergencies.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old
* ASA score of 1-3
* Elective or urgent surgery planned to last at least 30 minutes under general anesthesia with endotracheal intubation

Exclusion Criteria:

* Any contraindication to the use of SGA devices considered by the anesthesiologist (Uncontrolled gastro-eosophageal reflux, oropharyngeal pathology or gross deformation, etc.)
* Any contraindication to the drugs planned by the trial
* Pregnancy
* Severe or uncontrolled obstructive pulmonary disease
* Significant cervical spine anomaly

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Time for intubation | Through study completion, an average of half an hour (no follow-up required)
  This outcome corresponds to the time required to intubate with endotracheal tube (ET) through the supra-glottic airway device. The timer will be started when the flexible fiberoptic intubation scope is inserted in the SGA, and will be stopped when the air cuff of the ET is inflated inside the trachea and carbon dioxide (CO2) is obtained. This outcome will be assessed by the either the performer or second person responsible for data collection.

SECONDARY OUTCOMES:
Success of intubation on first attempt | Through study completion, an average of half an hour (no follow-up required)
  This outcome is dichotomic and represents success of intubation through the SGA on the first attempt. An attempt will be defined as any lowering of the ET towards the glottis. Thus, any raise of the ET to its original position on the fiberoptic intubation scope will be considered as a failed attempt. Similarly, any removal of the fiberoptic scope from the SGA will be considered as a failed attempt, regardless of an attempt to lower the ET. This primary outcome is dichotomous and answers to the question: "Was the first attempt successful?"
Success of intubation through the SGA | Through study completion, an average of half an hour (no follow-up required)
  Regardless of the number of attempts, this outcome will be considered positive if the ET penetrated the trachea, the air cuff was inflated and capnography is positive, sustained and with normal values. A failed intubation would be, for example, to leave the SGA in place for the whole surgery or to remove the SGA to complete the endotracheal intubation.
Number of attempts for intubation | Through study completion, an average of half an hour (no follow-up required)
  For example, the ET is lowered and does not enter the glottis, and is raised up again while the scope is removed from the SGA : "one" failed attempt will be noted. If the scope is entered in the SGA, no attempt to lower the ET and the scope is removed : "one" failed attempt will also be noted. However, if the scope is inserted in the SGA, the ET is lowered a first time and raised on the scope, and the ET is lowered a second time and raised again on the scope, "two" failed attempts will be considered.
Time for whole procedure | Through study completion, an average of half an hour (no follow-up required)
  The time for whole procedure corresponds to the sum of the time required for installation of the SGA device and the time required for intubation through the device.
Laryngeal view grades | Through study completion, an average of half an hour (no follow-up required)
  An evaluation of the laryngeal view on the first attempt of fibroscopy will be evaluated by the attending anesthesiologist with the following scale :
  * Grade 1 : whole vocal cords are seen, the epiglottis is not seen at all
  * Grade 2 : larynx plus the posterior surface of epiglottis are seen
  * Grade 3 : the anterior tip of the epiglottis is seen
  * Grade 4 : the anterior tip of the epiglottis is seen and encroaching on the view of vocal cords obstructing <50% of view
  * Grade 5 : the epiglottis is completely obstructing the SGA opening, no view is seen
Easiness of insertion and ventilation of the SGA | Through study completion, an average of half an hour (no follow-up required)
  The easiness of insertion and ventilation will be graded using the following scale, as proposed by Talaat and al. in his trial on Air-Q and Fastrach devices.
  * Easy means obtaining an effective airway, defined as normal chest movement and a square wave capnograph trace, from the first attempt
  * Moderate means obtaining an effective airway in the second or third attempt with some manipulation of the technique of insertion
  * Difficult means failure to obtain an effective airway after three attempts
Easiness of intubation | Through study completion, an average of half an hour (no follow-up required)
  The easiness of intubation will be subjectively evaluated by the attending anesthesiologist using the following scale:
  * Easy, meaning that railing the ET into the trachea was easy
  * Moderate, meaning that railing the ET needed mild corrective manoeuvers and the procedure was mildly longer than expected
  * Difficult, meaning that railing the ET was considerably longer than expected and that many corrective manœuvres were done, as removing and reinserting the fiberoptic scope.
Easiness of removal of the SGA after a completed endotracheal intubation | Through study completion, an average of half an hour (no follow-up required)
  The anesthesiologist will be asked to report a subjective evaluation of the removal of the SGA once the patient is intubated.
  * Easy removal
  * Moderate difficulty
  * Hard
  * Impossible
Adverse events | Through study completion, an average of half an hour (no follow-up required)
  The research team will report any adverse events. For example, accidental extubation during the removal of the SGA, blood on the device when removed, desaturation under 90%. As previously mentioned, if the attending anesthesiologist wants to stop the protocol for different reasons, as unsatisfactory ventilation, the standardized manipulations will be stopped and the anesthesiologist will pursue airway management according to his preferences.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-José Colas, MD, Principal Investigator — Centre Hospitalier Universitaire de Sherbrooke (CHUS)
Locations (1):
- Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Talaat AH, Mostafa AEE, Mohsen ME, Hesham SA. Comparative study between Air-Q and Intubating Laryngeal Mask Airway when used as conduit for fiber-optic. Egyptian Journal of Anaesthesia 30(2), 2013
- [Background] Apfelbaum JL, Hagberg CA, Caplan RA, Blitt CD, Connis RT, Nickinovich DG, Hagberg CA, Caplan RA, Benumof JL, Berry FA, Blitt CD, Bode RH, Cheney FW, Connis RT, Guidry OF, Nickinovich DG, Ovassapian A; American Society of Anesthesiologists Task Force on Management of the Difficult Airway. Practice guidelines for management of the difficult airway: an updated report by the American Society of Anesthesiologists Task Force on Management of the Difficult Airway. Anesthesiology. 2013 Feb;118(2):251-70. doi: 10.1097/ALN.0b013e31827773b2. No abstract available. PMID 23364566
- [Derived] Laferriere-Langlois P, Dion A, Guimond E, Nadeau F, Gagnon V, D'Aragon F, Sansoucy Y, Colas MJ. A randomized controlled trial comparing three supraglottic airway devices used as a conduit to facilitate tracheal intubation with flexible bronchoscopy. Can J Anaesth. 2023 May;70(5):851-860. doi: 10.1007/s12630-023-02444-z. Epub 2023 Apr 13. PMID 37055702